CLINICAL TRIAL: NCT04889157
Title: AN 8-WEEK, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED PHASE 1 STUDY TO EVALUATE THE PHARMACOKINETICS, PHARMACODYNAMICS, SAFETY AND TOLERABILITY OF PF-06882961 IN CHINESE ADULTS WITH TYPE 2 DIABETES MELLITUS
Brief Title: A Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of PF-06882961 in Chinese Adults With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C3421028
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — danuglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PF-06882961 (Experimental): Participants will be titrated up to 6 weeks of the 8-week dosing duration to reach desired dose level 120 mg
  Interventions: Drug: PF-06882961
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06882961 — Participants will be administered active doses, taking 3 tablets twice daily (BID) for 8 weeks except Day 1 (QD)
  Arms: PF-06882961
Drug: Placebo — 3 matching placebo tablets taken twice daily (BID) except Day 1 (QD)
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind (sponsor open), placebo controlled study in adult Chinese participants with T2DM who are receiving metformin as background antihyperglycemic medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM who are taking metformin monotherapy as their only antihyperglycemic treatment
* HbA1c greater than or equal to 7% and less than or equal to 10.5%
* Total body weight >50 kg (110 lb) with BMI of 22.5 to 45.4 kg/m^2

Exclusion Criteria:

* Any condition possibly affecting drug absorption
* Diagnosis of Type 1 diabetes mellitus or secondary forms of diabetes
* History of myocardial infarction, unstable angina, arterial revascularization, stroke, heart failure, or transient ischemic attack within 6 months of Screening
* Any malignancy not considered cured
* Personal or family history of MTC or MEN2, or participants with suspected MTC
* Acute pancreatitis or history of chronic pancreatitis
* Acute gallbladder disease
* Known history of HIV, hepatitis B, hepatitis C or syphilis, or positive testing of them
* Supine blood pressure greater than or equal to 160 mmHg (systolic) or greater than or equal to 100 mmHg (diastolic)
* Clinically relevant ECG abnormalities
* Positive urine drug test
* Clinical relevant laboratory tests abnormalities

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421028

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo BID (except QD in the morning on Day 1) from Days 1-56.
- PF-06882961 BID: Participants received PF-06882961 BID (except QD in the morning on Day 1) following dose titration schema: 10 mg on Days 1-7, 20 mg on Days 8-14, 40 mg on Days 15-21, 60 mg on Days 22-28, 80 mg on Days 29-35, 100 mg BID on Days 36-42, 120 mg from Days 43-56.
Period: BLINDED TREATMENT
Arm/Group | Placebo | PF-06882961 BID
Started | 5 | 15
Discontinued | 0 | 0
Completed | 5 | 15
Not Completed | 0 | 0
Period: Follow-Up
Arm/Group | Placebo | PF-06882961 BID
Started | 5 | 15
Received Treatment | 5 | 15
Completed | 5 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who were randomized and received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06882961 BID | Total
Number analyzed (Participants) | 5 | 15 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean (SD) | 50 (4.64) | 49.5 (7.22) | 49.6 (6.56)
Age, Customized [Number; unit: Participants]
  20-44 Years | 1 | 4 | 5
  45-60 Years | 4 | 11 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 9
  Male | 4 | 7 | 11
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 5 | 15 | 20
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic or Latino | 5 | 15 | 20

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to 24 Hours (AUC24) of PF-06882961 10 mg Single Dose on Day 1
Description: AUC24 is the area under the plasma concentration-time profile from time zero to the time 24 hours. The planned analysis was not considered reliable by the sponsor.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 10, 12, 14, 24 hours post dose on Day 1
Population: All participants randomized and treated with PF-06882961 who had at least 1 plasma concentration value collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliter (ng*hr/mL)
Groups:
- PF-06882961 10 mg Single Dose: Participants received single dose of PF-06882961 on Day 1.
Arm/Group | PF-06882961 10 mg Single Dose
Number analyzed (Participants) | 15
nanogram*hour per milliter (ng*hr/mL) | 287.4 (52)

2. Primary Outcome: Maximum Observed Concentration (Cmax) of PF-06882961 10 mg Single Dose on Day 1
Description: Cmax is the maximum observed plasma concentration over 24 hours. The planned analysis was not considered reliable by the sponsor.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 10, 12, 14, 24 hours post dose on Day 1
Population: All participants randomized and treated with PF-06882961 who had at least 1 plasma concentration value collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliter (ng/mL)
Groups:
- PF-06882961 BID: Participants received single dose of PF-06882961 on Day 1.
Arm/Group | PF-06882961 BID
Number analyzed (Participants) | 15
nanogram per milliter (ng/mL) | 37.37 (39)

3. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Supine blood pressure and pulse rate were measured with the participant's arm supported at the level of the heart and recorded to the nearest mmHg after approximately 5 minutes of rest and maximum absolute values and maximum changes from baseline from time-matched baseline were evaluated at the investigator's discretion.
Time Frame: Baseline up to 14 days after last dose (Day 70)
Population: All participants randomly assigned to study intervention and who had at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 BID
Number analyzed (Participants) | 5 | 15
Participants
  Supine systolic blood pressure (mmHg) change >=30 mm Hg increase | 1 | 3
  Supine systolic blood pressure (mmHg) change >=30 mm Hg decrease | 0 | 2
  Supine diastolic blood pressure (mmHg) change >=20 mm Hg increase | 1 | 6
  Supine diastolic blood pressure (mmHg) change >=20 mm Hg decrease | 0 | 1
  Supine pulse rate (beats per minute [bpm]) value >120 bpm | 0 | 1

4. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG)
Description: Standard 12-lead ECGs utilizing limb leads were collected using an ECG machine that automatically calculated the heart rate and measures PR, QT, and QT interval corrected for heart rate (QTc) and QRS complex.
Time Frame: Baseline up to 14 days after last dose (Day 70)
Population: All participants randomly assigned to study intervention and who had at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 BID
Number analyzed (Participants) | 5 | 15
Participants
  PR interval not otherwise specified (msec) %change >=50% | 0 | 1
  QTcF not otherwise specified (msec) 450 < Value <=480 | 1 | 1

5. Secondary Outcome: Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An serious adverse event was defined as any untoward medical occurrence that,at any dose:resulted in death;was life-threatening;required inpatient hospitalization or prolongation of existing hospitalization;resulted in persistent disability/incapacity; was a congenital anomaly/birth defect;or other serious situations such as important medical events. The investigator was required to use clinical judgment to assess the potential relationship between investigational product and each AE, to define an treatment-related AE.
Time Frame: Baseline up to 35 days after last dose (Day 91)
Population: All participants randomly assigned to study intervention and who had at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 BID
Number analyzed (Participants) | 5 | 15
Participants
  Participants with non-serious AEs | 5 | 14
  Participants with serious adverse events | 0 | 0

6. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory tests (including hematological, clinical chemistry, urinalysis tests) were reported and abnormality was determined at the investigator's discretion.
Time Frame: Baseline up to 14 days after last dose (Day 70)
Population: All participants randomly assigned to study intervention and who had at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06882961 BID
Number analyzed (Participants) | 5 | 15
Participants
  Hematology - Neutrophils (10^3/mm3) >1.2xupper limit of norma (ULN) | 0 | 1
  Hematology - Basophils (10^3/mm3) >1.2xULN | 0 | 1
  Chemistry - Urate (mg/dL) >1.2xULN | 0 | 4
  Chemistry - high-density lipoprotein cholesterol (mg/dL) <0.8xlower limit of normal (LLN) | 2 | 1
  Chemistry - Triglycerides (mg/dL) >1.3xULN | 0 | 3
  Chemistry - Thyrotropin (uIU/mL) <0.8xLLN | 0 | 1
  Chemistry - Bile Acid (umol/L) >1.0xULN | 0 | 1
  Urinalysis - Urine Glucose ≥1 | 3 | 6
  Urinalysis - Urine Ketones (Scalar) ≥1 | 0 | 2
  Urinalysis - Urine Protein ≥1 | 0 | 1
  Urinalysis - Urine Hemoglobin (Scalar) ≥1 | 1 | 3
  Urinalysis - Urine Urobilinogen ≥1 | 0 | 2
  Urinalysis - Urine Nitrite (Scalar) ≥1 | 0 | 1
  Urinalysis - Urine Leukocyte Esterase (Scalar) ≥1 | 0 | 2

7. Primary Outcome: AUC24 of PF-06882961 in Participants Received 40 mg BID, 80 mg BID, and 120 mg BID PF-06882961
Description: AUC24 was measured on Day 21, 35, and 56 for dose 40 mg BID, 80 mg BID, and 120 mg BID, respectively. The planned analysis was not considered reliable by the sponsor.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 10, 12, 14, 24 hours post dose on Day 21 (40 mg BID), 35 (80 mg BID), and 56 (120 mg BID)
Population: All participants randomized and treated with PF-06882961 who had at least 1 plasma concentration value collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- PF-06882961 40 mg BID; PF-06882961 80 mg BID; PF-06882961 120 mg BID: Participants received PF-06882961 BID (except QD in the morning on Day 1) following dose titration schema: 10 mg on Days 1-7, 20 mg on Days 8-14, 40 mg on Days 15-21, 60 mg on Days 22-28, 80 mg on Days 29-35, 100 mg BID on Days 36-42, 120 mg from Days 43-56.
Arm/Group | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 15 | 15 | 14
ng*hr/mL | 1446 (236) | 1012 (1414) | 984.9 (2327)

8. Primary Outcome: Maximum Observed Concentration, Steady State (Cmax,ss) of PF-06882961 in Participants Received 40 mg BID, 80 mg BID, and 120 mg BID PF-06882961
Description: Cmax,ss was measured on Day 21, 35, and 56 for dose 40 mg BID, 80 mg BID, and 120 mg BID, respectively. The planned analysis was not considered reliable by the sponsor.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 10, 12, 14, 24 hours post dose on Day 21 (40 mg BID), 35 (80 mg BID), and 56 (120 mg BID)
Population: All participants randomized and treated with PF-06882961 who had at least 1 plasma concentration value collected.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06882961 40 mg BID | PF-06882961 80 mg BID | PF-06882961 120 mg BID
Number analyzed (Participants) | 15 | 15 | 14
ng/mL | 150.3 (176) | 98.92 (1059) | 110.5 (3069)

ADVERSE EVENTS:
Time Frame: Baseline up to 35 days after last dose (Day 91)
Arm/Group | Placebo | PF-06882961 BID
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/15
Other Adverse Events (participants affected / at risk) | 5/5 | 14/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | PF-06882961 BID (N=15)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 2
Eye pain (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 12
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 12
Regurgitation (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 12
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Blood pressure increased (Investigations) | 0 | 2
Blood uric acid increased (Investigations) | 0 | 2
Hepatic enzyme increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 2 | 4
Sleep deficit (Nervous system disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
In this study, a Quality Event was identified upon review of the PK data after the final study database release. This Quality Event was identified as non-compliance to study intervention per retrospective investigation post database release. Due to the Quality Event, the PK results of the study were considered not reliable by the sponsor and should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT04889157/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT04889157/SAP_001.pdf